CLINICAL TRIAL: NCT01703273
Title: Structured Low-level Intervention vs. Treatment as Usual Evaluated in a Randomized Controlled Trial for Adolescents With Extreme Obesity, Subproject 2
Brief Title: Low-level Intervention for Adolescents With Extreme Obesity
Acronym: STEREO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Dr. Martin Wabitsch (Other)
Collaborators: University of Witten/Herdecke (Other); Charite University, Berlin, Germany (Other); University of Leipzig (Other); Universität Duisburg-Essen (Other); University of Ulm (Other); Zentrum für klinische Studien Essen (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. Martin Wabitsch, Prof. Dr. med, University of Ulm
Organization: University of Ulm (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: U1111-1131-4384b; DRKS00004195 (Registry Identifier: Deutsches Register Klinischer Studien); 01GI1120B (Other Grant/Funding Number: Bundesministerium für Bildung und Forschung)
Record Dates: First submitted 2012-08-07; First posted 2012-10-10 (Estimated); Last update posted 2018-06-13 (Actual); Status verified 2018-06

CONDITIONS: Obesity; Extreme Obesity
Keywords: Extreme Obesity Keywords: obesity, adiposity, psychosocial, healthcare, co-morbidities, low key intervention, quality of life
MeSH Terms: conditions — Obesity; Obesity, Morbid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- low key intervention (Experimental)
  Interventions: Behavioral: manual based low key group intervention (innovation)
- routine care (Active Comparator)
  Interventions: Behavioral: standardized, manual based routine care

INTERVENTIONS:
Behavioral: manual based low key group intervention (innovation) — 6 sessions offered over the course of 3-6 months focus on improvement of quality of life and psychosocial functioning . Topics covered are: 1) social competencies, 2) body image, 3) coping with mobbing and anger, 4) coping with stress, 5) life satisfaction, and 6) psychological well being. The planned intervention does not primarily focus on weight loss.
  Arms: low key intervention
Behavioral: standardized, manual based routine care — 6 sessions offered over the course of 3-6 months with a focus on weight loss. The topics 1) causes, consequences and treatment options of obesity, 2) nutrition, 3) eating behaviors and problem solving strategies, 4) self esteem and emotional eating, 5) exercise, and 6) use of media, will be covered.
  Arms: routine care

SUMMARY:
While adolescents with obesity and extreme obesity are at increased risk for health complications, especially adolescents with extreme obesity rarely seek medical care, and sustained weigh loss is hardly ever achieved. One of the underlying reasons might be the lack of adequate treatment options.

In this multicenter study, we aim to test a new, low key group intervention focusing on improving compliance and psychosocial functioning. The study is a subproject of the Medical and psychosocial implications of adolescent extreme obesity - acceptance and effects of structured care, short: "Youth with Extreme obesity Study (YES)", which aims at improving the medical care and social support structures for youth with obesity and extreme obesity in Germany.

Obese youth and young adults (BMI ≥ 30kg/m2) between the ages of 14 and 24.9 years (initially up to 21 years) are eligible to participate. Participants will be asked to complete a series of questionnaires on their general health, psychosocial situation and wellbeing, and will be offered a thorough medical evaluation. Individuals who complete the baseline evaluations will be invited to participate in 6 group sessions over a 3 months period. Group assignment to the psycho-social intervention vs. routine care group will be at random, like throwing a dice. After 6 months, participants will complete further questionnaires to evaluate the effects of the interventions on quality of life and psycho-social functionning.

The study will show the acceptance and effectiveness of a new intervention focusing on improving compliance and psychosocial functioning in adolescents with extreme obesity, and thereby inform the development of new treatment and support options for these adolescents. If interested, participants are invited to participate in additional components of YES, and to receive medical care and psycho-social support.

DETAILED DESCRIPTION:
While obese youth are at high risk for co-morbidities, especially the extremely obese individuals rarely seek medical care. The underlying reasons are poorly understood, but patient inherent factors and the lack of adequate treatment options may play a role.

In this multicenter study, we aim to assess the acceptance and effectiveness of a manual based low key group intervention focusing on improving compliance and psychosocial functioning in adolescents with morbid obesity (BMI≥35kg/m2), in comparison to routine care. Youth with more moderate degrees of obesity (BMI 30-34.9kg/m2) will serve as an additional control group. The study is part of the Medical and psychosocial implications of adolescent extreme obesity - acceptance and effects of structured care", short: "Youth with extreme obesity Study (YES), which also comprises the recruitment and characterization of obese (BMI 30-34.9kg/m2) and extremely obese (BMI ≥ 35kg/m2) youth from different healthcare- and non healthcare settings, a structured prospective evaluation of adolescent bariatric surgery, economic assessments of the financial burden of extreme adolescent obesity on the healthcare system, and a long-term prospective observation study.

Based on the current state of knowledge, we will test the a priori ordered hirarchy of hypotheses:

1. The compliance rate 6 months after randomization is higher in subjects in the low key intervention group compared to the standard care group.
2. Covariant-adjusted changes in quality of life (assessed by DISABKIDS scale) between baseline and the 6 months follow up will be more pronounced in the low key intervention group compared to the standard care group.

The five participating university centers are distributed across 4 geographic regions in the North (Berlin), in the West (Essen/Datteln), in the East (Leipzig) and in the South (Ulm) of Germany, and will therefore render data that are representative of Germany as a whole. We will screen a 600 adolescents age 14 to 24.9 years (initially up to 21 years; this was changed in an amendment in February 2013) with extreme obesity (BMI ≥ 35 kg/m2) and 600 adolescents with obesity (BMI 30-34.9 kg/m2) over a 24 months period. A total of 350 subjects will be enrolled. Baseline assessments include an array of standardized questionnaires and validated instruments to assess health, psycho-social situation, psychiatric co-morbidities and health related quality of life, as well as an in-depth medical evaluation. Individuals who complete the baseline evaluations will be invited to participate in 6 group sessions over a 3 months period. Group assignment to the low key intervention vs. standard care group will be at random. The effects of the interventions on health related quality of life and psycho-social functioning will be assessed via questionnaires after 6 months. Subsequently, subjects will be invited to participate in additional components of YES.

The project will reveal the effectiveness and safety of a manual based low key group intervention focusing on improving compliance and psychosocial functioning in adolescents with morbid obesity, and thereby inform the development of new treatment and support options for these adolescents in Germany.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥30kg/m2
* sufficient German language skills

Exclusion Criteria:

* Circumstances that require immediate inpatient care (e.g. severe somatic or psychiatric illness)
* obvious cognitive disability

Ages: 14 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 119 (Actual)
Dates: Start 2012-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Composite primary endpoint (tested hierarchically) of a) compliance rate and b) changes in health related quality of life. | baseline and 6 months
  a) Number of regular participants at 6 months follow up will be divided by number of participants at baseline. b) Changes (randomization - 6 months follow up) in the 37 item DISABKIDS questionnaire will be assessed.

SECONDARY OUTCOMES:
Changes in the 6 subscales of DISABKIDS | baseline and 6 months
  The 37 item DISABKIDS questionnaire will be applied twice, and the score difference in each of the 6 subscales will be calculated for each subject.
Changes in quality of life | baseline and 6 months
  The 52 item KIDSCREEN-52 questionnaire will be applied twice, and the score difference will be calculated for each subject.
Changes in self-esteem | baseline and 6 months
  The Rosenberg's scale patient questionnaire will be applied twice, and the score difference will be calculated for each subject.
Changes in self reported time spent outside the home | baseline and 6 months
  The time spent outside the home will be elicited twice via standardized patient questionnaire (modified after KIGGS and TeenLABS), and the time difference will be calculated for each subject.
Changes in depression symptoms | baseline and 6 months
  The Becks Depression Inventory 2 questionnaire will be applied twice, and the score difference will be calculated for each subject. Answers will be reviewed immediately to identify and treat subjects at risk for self harm.
Changes in perceived stress | baseline and 6 months
  The Fliege scale questionnaire will be applied twice, and the score difference will be calculated for each subject.
Changes in the self reported attendance of school, apprenticeship, or work | baseline and 6 months
  The attendance of school, apprenticeship, or work will be elicited twice via standardized patient questionnaire (modified after KIGGS and TeenLABS), and the time difference will be calculated for each subject.
Changes in self reported physician- / and therapist contacts | baseline and 6 months
  Physician- / and therapist contacts will be elicited twice via standardized patient questionnaire (modified after KIGGS and TeenLABS), and the difference will be calculated for each subject.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Wabitsch, Prof. Dr. med., Principal Investigator — University of Ulm; Susanna Wiegand, Dr. med., Principal Investigator — Charite University, Berlin, Germany; Thomas Reinehr, Prof. Dr. med., Principal Investigator — University of Witten/Herdecke; Johannes Hebebrand, Prof. Dr. med., Study Chair — Universität Duisburg-Essen; Wieland Kiess, Prof. Dr. med., Principal Investigator — University of Leipzig
Locations (6):
- Germany (6):
  - Ambulatory Obesity Program, Charité University, Berlin, Berlin
  - Vestische Kinderklinik, University of Witten/Herdecke, Datteln
  - Center for Clinical Trials Essen, Essen
  - University Duisburg-Essen, Essen
  - University Hospital Leipzig, Leipzig
  - Dept for Pediatrics and Adolescent Medicine, University of Ulm: Interdisciplinary obesity clinic, Ulm

REFERENCES:
- [Derived] Muhlig Y, Scherag A, Bickenbach A, Giesen U, Holl R, Holle R, Kiess W, Lennerz B, Lutke Brintrup D, Moss A, Neef M, Ose C, Reinehr T, Teuner CM, Wiegand S, Wolters B, Wabitsch M, Hebebrand J. A Structured, Manual-Based Low-Level Intervention vs. Treatment as Usual Evaluated in a Randomized Controlled Trial for Adolescents with Extreme Obesity - the STEREO Trial. Obes Facts. 2017;10(4):341-352. doi: 10.1159/000475717. Epub 2017 Aug 9. PMID 28787738
- [Derived] Wabitsch M, Moss A, Reinehr T, Wiegand S, Kiess W, Scherag A, Holl R, Holle R, Hebebrand J. Medical and psychosocial implications of adolescent extreme obesity - acceptance and effects of structured care, short: Youth with Extreme Obesity Study (YES). BMC Public Health. 2013 Aug 29;13:789. doi: 10.1186/1471-2458-13-789. PMID 23987123
- See also: study homepage — http://www.adipositasforschung-ulm.de/index.php?id=69